CLINICAL TRIAL: NCT05253729
Title: Efficacy of Focused Shockwave Therapy in Patients With Moderate to Severe Carpal Tunnel Syndrome, a Single-blinded Randomized Controlled Trial
Brief Title: Efficacy of Focused Shockwave Therapy in Patients With CTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MURA 2017/708
Record Dates: First submitted 2022-01-24; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome, ESWT, shockwave therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focused Extracorporeal Shock Wave Therapy (F-ESWT) (Experimental): Participants in the intervention group received low-intensity F-ESWT once a week for three sessions plus conservative treatment.
  Interventions: Device: Focused ESWT
- Control (Active Comparator): Participants in the control group received only conservative treatment including disease education, advice about proper posture and activity, night wrist splint and nerve gliding exercise.
  Interventions: Behavioral: Control

INTERVENTIONS:
Device: Focused ESWT — F-ESWT (dose 0.01-0.15 mJ/mm2, frequency 4-5 Hz, 1500 shocks) was applied perpendicular to the palmar side of the wrist which was done once a week for a total of three sessions plus conservative treatment.
  Other Names: F-ESWT
  Arms: Focused Extracorporeal Shock Wave Therapy (F-ESWT)
Behavioral: Control — Participants in the control group received only conservative treatment including disease education, advice about proper posture and activity, night wrist splint and nerve gliding exercise.
  Arms: Control

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common entrapment of upper extremity. Patients with CTS will experience symptoms of pain, numbness of tingling sensation along the median nerve distribution. In more severe case, patients may have difficult manipulating objects that disturb function and patient's quality of life. Extracorporeal Shockwave Therapy (ESWT) is one of physical modalities that uses to treat many musculoskeletal disorders. For CTS, previous evidence showed that ESWT can improve symptoms, function as well as electrophysiologic parameters. However, standardized guidelines as well as the study in patients with moderate to severe CTS has not been established. Thus, the objective of the present study was to evaluate efficacy of ESWT in term of symptoms, function, electrophysiologic parameters, as well as sonography of median nerve in patients with moderate to severe CTS.

DETAILED DESCRIPTION:
* The present study was a single-blinded randomized controlled trial comparing the efficacy of focused ESWT (F-ESWT) to conservative treatment in patients with CTS.
* 24 patients who was diagnosed as CTS based on symptoms of CTS and physical examination. They were randomly allocated into two groups (21 patients per group), mainly F-ESWT plus conservative treatment and conservative treatment only.
* Outcome measures were BCTQ including symptom and function subscales, electrophysiologic parameters, and sonography to evaluate cross-sectional area (CSA) of the median nerve. All measures were recorded at baseline, 3 weeks and 6 weeks of treatment.
* Statistical analysis was performed to determine changes within the same group and compare difference between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who were diagnosed as CTS based on the American Academy of neurology
2. Participants who have electrodiagnostic evidence of CTS according to American Association of Neuromuscular and Electrodiagnostic Medicine (AANEM) guidelines for diagnosis of CTS. The severity of median nerve compression at wrist was moderate to severe degree.
3. Patients who were not treated by NSAIDs within 2 weeks prior to participating in the study.

Exclusion Criteria: The below exclusion criteria were applied only on the affected hand that were enrolled to the study

1. History of previous carpal tunnel release.
2. Receiving steroid injections for the treatment of CTS
3. History of infection or severe inflammation on the wrist
4. Contraindications for focused ESWT, such as arrhythmias, pacemakers, bleeding disorders, pregnancy, severe osteoporosis, and cancer.
5. Participants who refused or requested withdrawal from the study.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Thai version of Boston Carpal Tunnel Questionnaire (T-BCTQ) | BCTQs and BCTQf were assessed changes from baseline to at 6 weeks of treatment.
  T-BCTQ was used to assess symptom severity and hand function in patients with CTS. This questionnaire consists of two parts, mainly BCTQ symptom severity (BCTQs) and BCTQ functional status (BCTQf). Total questions for each part were 11 and 8 questions, respectively with scores raging from 1-5.

SECONDARY OUTCOMES:
Electrodiagnostic parameters: Distal Sensory Latency (DSL) | Changes of DSL was assessed from baseline to at 6 weeks of treatment.
  DSL was evaluated using Cadwell Sierra Summit model IEC601-1.
Electrodiagnostic parameters: Distal Motor Latency (DML) | Changes of DSL was assessed from baseline to at 6 weeks of treatment.
  DML was evaluated using Cadwell Sierra Summit model IEC601-1.
Electrodiagnostic parameters: Sensory Nerve Action Potential (SNAP) amplitude | SNAP amplitude was assessed from baseline to at 6 weeks of treatment.
  Sensory nerve action potential (SNAP) amplitude was evaluated using Cadwell Sierra Summit model IEC601-1.
Electrodiagnostic parameters: Compound Muscle Action Potential (CMAP) amplitude | Changes of CMAP amplitude was assessed from baseline to at 6 weeks of treatment.
  CMAP amplitude was evaluated using Cadwell Sierra Summit model IEC601-1.
Electrodiagnostic parameters: Total area under curve (TAUC) | Changes of TAUC was assessed from baseline to at 6 weeks of treatment.
  TAUC was evalauted using Cadwell Sierra Summit model IEC601-1.

OTHER OUTCOMES:
Median nerve cross-sectional area (CSA) at wrist level | Changes of median nerve CSA at wrist were assessed from baseline to at 6 weeks of treatment.
  Median nerve CSA at wrist (pisiform level) was assessed by ultrasonography.
Median nerve cross-sectional area (CSA); wrist to forearm ratio | Median nerve CSA (wrist to forearm ratio) were assessed changes from baseline to at 6 weeks of treatment.
  Median nerve CSA was assessed by ultrasonography in two levels, mainly at pisiform level and at the level of pronator quadratus muscle. CSA were then determined for wrist to forearm ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Punpetch Siriratna, MD, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Punpetch Siriratna, Bangkok, Thailand